CLINICAL TRIAL: NCT06346366
Title: Glucose Control Through a Bihormonal Artificial Pancreas in Patients After Total Pancreatectomy (PANORAMA): Randomized Controlled Crossover Trial
Brief Title: Glucose Control Through a Bihormonal Artificial Pancreas in Patients After Total Pancreatectomy
Acronym: PANORAMA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, M.G. Besselink, Marc Besselink, Prof. Dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NL.82557.018.22
Record Dates: First submitted 2024-02-22; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Pancreatic Neoplasms; Type 3c Diabetes; Total Pancreatectomy
Keywords: Bihormonal artificial pancreas
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients are randomized to a 3-month treatment period with the bihormonal artificial pancreas (BIHAP) (preceded by a training period) or a 3-month treatment with their current diabetes care. Hereafter, all patients will cross over.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open loop (Active Comparator): The control arm (open loop) consists of standard treatment for diabetes with continuous subcutaneous insulin infusion or insulin injections for 3 months.
  Interventions: Device: Bihormonal artificial pancreas (BIHAP) / closed loop
- Closed loop (Experimental): The intervention arm is 3 months closed loop control of blood glucose with the BIHAP. The BIHAP contains a self-learning algorithm which automatically maintains the glucose levels within target limits via subcutaneous administration of insulin (Humalog®) and glucagon. Patients complete a training period before the intervention period will start.
  Interventions: Device: Bihormonal artificial pancreas (BIHAP) / closed loop

INTERVENTIONS:
Device: Bihormonal artificial pancreas (BIHAP) / closed loop — The investigational device is a dual-hormonal fully closed loop system (BIHAP; industrial name AP® 5, Inreda Diabetic B.V.) which aims at optimally controlling plasma glucose levels. This BIHAP contains of two pumps for subcutaneous infusion of either insulin (Humalog, 3 ml pre-fill cartridge, Eli Lilly) or glucagon (GlucaGen, Novo Nordisk; 3.15 ml cartridge Accu-Chek Spirit, Roche) via an infusion set (Accu-Chek Insight Flex or AccuChek Flex Link, Roche), two subcutaneously placed glucose-sensors (Guardian, Medtronic) and an algorithm driving pump infusion rates based on the sensor input. Daily self-measurements of blood glucose (SMBGs; Accu-Chek Instant, Roche) are needed for calibration of the glucose sensors.
  The BIHAP-system has to be worn continuously, except while showering.
  Other Names: Current regular diabetes treatment / open loop

SUMMARY:
In recent years total pancreatectomy is increasingly performed in selected patients due to the increasing use of preoperative chemotherapy, making more patients operable. After total pancreatectomy, all patients develop insulin dependent diabetes mellitus (IDDM). Glucose control in these patients is challenging due to the complete absence of both pancreatic insulin and glucagon secretion, and most patients report decreased quality of life due to fear of hypoglycemic events and the need for continuous glucose monitoring.

The CE marked bihormonal artificial pancreas (BIHAP) provides continuous fully automatic glucose monitoring and administration of insulin and glucagon using a self-learning algorithm. In a recent pilot study (APPEL5+, NL.8871) the BIHAP was being compared to current diabetes treatment in 10 patients after total pancreatectomy. This trial demonstrated that treatment with BIHAP was safe and improved time spent in euglycemia significantly during one week treatment (78.30%, [IQR 71.05%-82.61%] vs. 57.38% [IQR 52.38%-81.35%], p=0.03).

Now, larger randomized studies with a longer treatment period are necessary to confirm safety and efficacy of BIHAP for the treatment of diabetes in patients after total pancreatectomy, with sufficient attention for long-term glycemic control (HbA1c) and patient-reported outcomes.

The PANORAMA trial will evaluate the efficacy of a 3-month treatment with BIHAP in 40 patients after total pancreatectomy as compared to a 3-month treatment period with current diabetes care in a randomized cross-over trial. Patients will be randomized to start with the BIHAP (after a training period) or current diabetes care (i.e. insulin pen or pump). Hereafter, all patients will cross over.

DETAILED DESCRIPTION:
Rationale:

Insulin dependent diabetes after total pancreatectomy (TP) is difficult to manage due to the complete absence of alfa and beta cells. In a recent pilot study in 10 patients after total pancreatectomy, treatment with a bihormonal closed loop system was safe and resulted in better glucose control compared to current open loop therapy.

Objective:

To assess the efficacy of a 3-month treatment with a bihormonal artificial pancreas (BIHAP) in patients after total pancreatectomy compared to current diabetes care.

Secondary objectives are to assess the safety of BIHAP treatment; quality of life during BIHAP treatment and additional efficacy parameters.

Study design:

PANORAMA is a randomized, cross-over trial performed in an outpatient setting comparing closed loop diabetes treatment with BIHAP to open loop with current diabetes care (i.e., insulin pump or pen therapy) in 40 adults after TP. Patients will be recruited from Dutch Pancreatic Cancer Group hospitals and randomized to a 3-month treatment period with the BIHAP (preceded by a 5-day training period) or a 3-month treatment with their current diabetes care. Hereafter, all 40 patients will cross over. Study population: This trial will comprise in total 40 adult patients with insulin dependent diabetes at least three months after total pancreatectomy.

Intervention: The intervention is 3 months closed loop control of blood glucose with the BIHAP. Patients complete a 5-day training period before the intervention period will start. The BIHAP contains a self-learning algorithm which automatically maintains the glucose levels within target limits via subcutaneous administration of insulin (Humalog®) and glucagon. The control arm (open loop) consists of standard treatment for diabetes with continuous subcutaneous insulin infusion or insulin injections for 3 months. After a wash-out period of 3 months, all patients will crossover to the other study arm.

Main study parameters/endpoints:

The primary endpoint will be time (in %) spent in the normal glucose range (3.9 mmol/l - 10.0 mmol/l).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

Patients will have to wear the prototype with two subcutaneous sensors and infusion sets continuously. There are no major risks associated with this study. The most prominent risk is failure of the BIHAP to regulate the plasma glucose concentration properly, which can result in hypo- or hyperglycemia. This may be caused by failure of the algorithm, technical failure or due to incorrect glucose measurements. However, with multiple risk control measures the risk for the patients is minimized. The system comprises a controller, a separate safety processor, as well as multiple alerts that are built in the system.

The potential benefits for each patient include a significantly better glycemic control, as well as improved quality of life because the BIHAP system completely takes over the glucose regulation, thereby minimizing the burden of life with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Age ≥18 years
* Insulin dependent diabetes after total pancreatectomy (patients who previously participated in APPEL 5+ are allowed to be included)
* At least three months after total pancreatectomy
* Patients using flash or continuous glucose sensor (Free Style Libre, Guardian or Medtronic) ,willing to scan this sensor at least three times per day during the control period and to remove this sensor during BIHAP treatment
* Undergoing treatment with CSII or subcutaneous insulin injections.

Exclusion Criteria:

* Known or suspected allergy to trial product(s) or related products;
* Suboptimal clinical condition, for instance due to active postoperative surgical complications, including skin condition prohibiting needle insertion;
* Actively participating in an investigational study (drug or device) wherein he/she has received treatment from an investigational study drug or device in the last 2 weeks before enrolment into this study, as per investigator judgment;
* Donation of blood or plasma in the past month, or in excess of 500 mL within 12 weeks prior to screening for other clinical trial related purposes;
* Current treatment with chemotherapy or when used less than 3 months prior to screening;
* BMI > 35 kg/m2;
* HbA1c > 97 mmol/ml (=11.0 %);
* Use of oral glucose-lowering medication;
* Limited ability to see, and to hear or feel alarms signals of the BIHAP;
* Use of acetaminophen (paracetamol) during the use of the BIHAP, as this may influence the sensor glucose measurements.
* Current pregnancy, breast feeding or planning to become pregnant during the trial or using ineffective birth control methods;
* Patients with a concomitant disease affecting metabolic control;
* Presence of a medical or psychiatric condition, longstanding serious adherence problems, anticipated problems in handing over diabetes control to a device or use of a medication that, in the judgment of the investigator, clinical protocol chair, or medical monitor, could compromise the results of the study or the safety of the participant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-04-25 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Time in range | During open and closed loop treatment (both 3 months)
  Time spent in euglycemia (glucose value 3.9-10.0 mmol/l or 70-180mg/dL) during BIHAP treatment

SECONDARY OUTCOMES:
Efficacy of open and closed loop system | During open and closed loop treatment (both 3 months)
  Additional metrics relating to glucose control will be compared between intervention and control period to provide more information about the efficacy of the BIHAP. This includes the following;
  * Day, night, and overall time spent in the following hypo-, and hyperglycemic ranges (percentage of time)
  * Percentage of time spent in the following categories:
    * Hypoglycemia level 1: <3.9 mmol/l;
    * Hypoglycemia level 2: <3.0 mmol/l;
    * Hyperglycemia level 1: >10mmol/l;
    * Hyperglycemia level 2: >13.9mmol/l.
Efficacy of open and closed loop system | During open and closed loop treatment (both 3 months)
  Additional metrics relating to glucose control will be compared between intervention and control period to provide more information about the efficacy of the BIHAP. This includes the following;
  - Glycemic, variability assessed by SD and CV (Coefficient of Variation)
Efficacy of open and closed loop system | During open and closed loop treatment (both 3 months)
  Additional metrics relating to glucose control will be compared between intervention and control period to provide more information about the efficacy of the BIHAP. This includes the following;
  - Daily insulin and glucagon use (in IE)
Efficacy of open and closed loop system | During open and closed loop treatment (both 3 months)
  Additional metrics relating to glucose control will be compared between intervention and control period to provide more information about the efficacy of the BIHAP. This includes the following;
  * Day, night and overall median sensor glucose concentration (mmol/l)
  * Median sensor glucose concentrations (mmol/l)
  * Mean HbA1c (mmol/ml)
Efficacy of open and closed loop system | During open and closed loop treatment (both 3 months)
  Additional metrics relating to glucose control will be compared between intervention and control period to provide more information about the efficacy of the BIHAP. This includes the following;
  - Percentage of patients achieving HbA1c ≤ 53 mmol/mol at baseline and after each treatment period
Adverse events and device issues associated with closed loop system with BIHAP | During open and closed loop treatment (both 3 months)
  Safety of glucose control with BIHAP treatment will be evaluated by assessing the incidence of (severe) adverse events and the incidence of device issues.
Patient reported outcomes on quality of life - WHO-5 | During open and closed loop treatment (both 3 months)
  To assess the impact of novel treatment with BIHAP on quality of life. The following questionnaires will be used to assess and compare quality of life during BIHAP treatment and regular treatment. All questionnaires will be filled at baseline, the start and end of both treatment arms;
  - World Health Organization-Five Well-Being Index (WHO-5) score; The total raw score, ranging from 0 to 25, is multiplied by 4 to give the final score, with 0 representing the worst imaginable well-being and 100 representing the best imaginable well-being.
Patient reported outcomes on quality of life - EQ-5D-5L | During open and closed loop treatment (both 3 months)
  To assess the impact of novel treatment with BIHAP on quality of life. The following questionnaires will be used to assess and compare quality of life during BIHAP treatment and regular treatment. All questionnaires will be filled at baseline, the start and end of both treatment arms;
  - Health-related quality of life scores (EQ-5D-5L); Overall current health is scored on a scale from 0-100, whereby 100 is labelled as 'The best health you can imagine' and 0 as 'The worst health you can imagine.
Patient reported outcomes on quality of life - DTSQc andDTSQs | During open and closed loop treatment (both 3 months)
  To assess the impact of novel treatment with BIHAP on quality of life. The following questionnaires will be used to assess and compare quality of life during BIHAP treatment and regular treatment. All questionnaires will be filled at baseline, the start and end of both treatment arms;
  - Diabetes Treatment and Satisfaction Questionnaire status and change (DTSQ-s and DTSQ-c) scores; The DTSQ status (DTSQs) items are scored on a scale from 6 to 0 and DTSQ change (DTSQc) items are on a scale from 3 to -3. The scale total is computed by adding the six items 1, 4, 5, 6, 7 and 8 to produce the Treatment Satisfaction scale total, which has a minimum of zero and a maximum of 36 on the DTSQs and a minimum of -18 and a maximum of 18 on the DTSQc.
Patient reported outcomes on quality of life - PAID-20 | During open and closed loop treatment (both 3 months)
  To assess the impact of novel treatment with BIHAP on quality of life. The following questionnaires will be used to assess and compare quality of life during BIHAP treatment and regular treatment. All questionnaires will be filled at baseline, the start and end of both treatment arms;
  - Problem Areas In Diabetes (PAID-20) score; PAID is a self-administered 20-item scale. Each item is scored from 0 (not a problem) to 4 (serious problem). The sum of all item scores multiplied by 1.25 gives the total PAID score, which ranges from 0 to 100, higher scores reflecting greater emotional distress. A score of 40 or above is indicative of severe emotional distress.
Patient reported outcomes on quality of life - HFS-II | During open and closed loop treatment (both 3 months)
  To assess the impact of novel treatment with BIHAP on quality of life. The following questionnaires will be used to assess and compare quality of life during BIHAP treatment and regular treatment. All questionnaires will be filled at baseline, the start and end of both treatment arms;
  - Hypoglycaemia Fear Survey-II (HFS-II) Worry subscale score; The HFS-II subscale scores and total score are sum scores of all or relevant subset of items ranging 0-60, 0-72, and 0-132 for the HFS-B, HFS-W, and HFS-II, respectively. Higher scores indicate higher fear of hypoglycemia.
Patient reported outcomes on quality of life - PSQI | During open and closed loop treatment (both 3 months)
  To assess the impact of novel treatment with BIHAP on quality of life. The following questionnaires will be used to assess and compare quality of life during BIHAP treatment and regular treatment. All questionnaires will be filled at baseline, the start and end of both treatment arms;
  - Pittsburg Sleep Quality Index score (PSQI); In scoring the PSQI, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Patient reported outcomes on quality of life - INSPIRE | During open and closed loop treatment (both 3 months)
  To assess the impact of novel treatment with BIHAP on quality of life. The following questionnaires will be used to assess and compare quality of life during BIHAP treatment and regular treatment. All questionnaires will be filled at baseline, the start and end of both treatment arms;
  - Insulin delivery systems: perceptions, ideas, reflections and expectations (INSPIRE) scores; The five response options are scored as 4 = Strongly Agree, 3 = Agree, 2 = Neither Agree or Disagree, 1 = Disagree, and 0 = Strongly Disagree. All items are responded to on this same scale and there are no reverse-scored items. Multiply the mean score calculated in step two by 25. This score represents a scaled score from 0 to 100 and was done in order to provide similar scaling as other commonly used quality of life scales. This final score will range from 0 to 100. Higher scores indicate more positive appraisal of automated insulin dosing
Patient reported outcomes on quality of life - Hypoglycaemia unawareness | During open and closed loop treatment (both 3 months)
  To assess the impact of novel treatment with BIHAP on quality of life. The following questionnaires will be used to assess and compare quality of life during BIHAP treatment and regular treatment. All questionnaires will be filled at baseline, the start and end of both treatment arms;
  - Hypoglycaemia unawareness (Gold-Clarke); Each question's response corresponds to "aware" (value 0) or "unaware" (value 1); scores are then summed. Scores of 0-2 are categorized as "aware", 4-7 as "unaware", and 3 as "indeterminant". The Gold questionnaire has only 1 question: "Do you know when your hypoglycemic episodes are commencing?" and is scored on a 7-point Likert scale. Scores of 1-2 are categorized as "Aware", 4-7 as "unaware", and 3 as "indeterminant".
Patient reported outcomes on quality of life - benefits and disadvantages of BIHAP treatment | During open and closed loop treatment (both 3 months)
  To assess the impact of novel treatment with BIHAP on quality of life. The following questionnaires will be used to assess and compare quality of life during BIHAP treatment and regular treatment. All questionnaires will be filled at baseline, the start and end of both treatment arms;
  - Patient reported benefits and disadvantages of BIHAP treatment, including continuation of BIHAP treatment if this was possible

OTHER OUTCOMES:
Other treatment endpoints - daily insulin and glucagon use | During open and closed loop treatment (both 3 months)
  - Insulin and glucagon use during the study at baseline and during each month for both treatment arms;
Other treatment endpoints - activity of BIHAP algorithm | During open and closed loop treatment (both 3 months)
  - The time that the control algorithm of the BIHAP is active. This will be given as mean with standard deviation or as median with IQR;
Other treatment endpoints - daily insulin use | During open and closed loop treatment (both 3 months)
  - Patient reported daily insulin use in the control group at 1, 2 and 3 months.
Other treatment endpoints - treatment related actions | During open and closed loop treatment (both 3 months)
  - Number of treatment related actions:
  * During BIHAP: number of hypoglycemic events, number of inserting new glucagon and/or insulin infusion sets and sensors, BIHAP alarm frequency, minor hazard frequency;
  * During the control period: number of hypoglycemic events, number of daily injections.
Other treatment endpoints - demographics | During open and closed loop treatment (both 3 months)
  * Demographic variables at baseline;
  * Concomitant medication use at baseline, an during each month for both treatment arms.
Other treatment endpoints - demographics | During open and closed loop treatment (both 3 months)
  - Demographic variables at baseline;
Other treatment endpoints - concomitant medication | During open and closed loop treatment (both 3 months)
  - Concomitant medication use at baseline, an during each month for both treatment arms.

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, Amsterdam, Netherlands